CLINICAL TRIAL: NCT06510816
Title: A Phase 3, Multicenter, Randomized, Parallel-Group, Double-Masked, 2-Arm, Sham Controlled Study of the Efficacy, Safety, and Tolerability of ANX007 Administered by Intravitreal Injection in Patients With Geographic Atrophy (GA) Secondary to Age Related Macular Degeneration (AMD)
Brief Title: A Study Investigating the Efficacy and Safety of Intravitreal (IVT) Injections of Vonaprument (Formerly ANX007) in Participants With Geographic Atrophy (GA)
Acronym: ARCHER II
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANX007-GA-02; 2024-515022-88-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Double-masked
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vonaprument (Experimental): Participants will receive vonaprument IVT injections every month during the 24-month treatment period.
  Interventions: Drug: Vonaprument
- Sham Group (Sham Comparator): Participants will receive Sham IVT injections every month during the 24-month treatment period.
  Interventions: Other: Sham Administration

INTERVENTIONS:
Drug: Vonaprument — Form: solution for injection; Route of Administration: IVT injection
  Other Names: ANX007
  Arms: Vonaprument
Other: Sham Administration — Form and Route of Administration: to mimic IVT injection (includes placement of the blunt opening of an empty, needleless syringe barrel on the conjunctiva in the inferotemporal quadrant of the eyeball to stimulate the pressure of an injection).
  Arms: Sham Group

SUMMARY:
The primary purpose of the study is to determine if IVT injections of vonaprument every month reduce vision loss in participants with GA secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GA of the macula secondary to AMD as determined by the Investigator and confirmed by the independent Central Reading Center.

Exclusion Criteria:

* Geographic atrophy due to other causes than AMD such as Stargardt disease, cone-rod dystrophy, pathologic myopia, or toxic maculopathies (for example, plaquenil maculopathy) in either eye.

NOTE: Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 659 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing a best corrected visual acuity (BCVA) ≥15-letter loss from baseline through the primary timepoint as assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) chart at any two consecutive visits. | The primary timepoint is based on accumulation of the target event rate, but no earlier than Month 12 and no later than Month 18

SECONDARY OUTCOMES:
Change From Baseline in the Hazard of ≥15 letter BCVA Loss Through Month 12 and Month 24 | Baseline, Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Annexon, Inc.
Locations (130):
- United States (70):
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - RCOC Clinical Research Institute Inc, Fullerton, California
  - Global Research Management, Glendale, California
  - Retina Consultants Medical Group, Modesto, California
  - Northern California Retina Vitreous Associates Medical Group, Inc., Mountain View, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Macula Retina Vitreous Research Institute, Torrance, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - RSC Research, LLC, Denver, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Retina Institute, Orlando, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Group of Florida, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Retina Associates - Elmhurst Location, Elmhurst, Illinois
  - University Retina, Oak Forest, Illinois
  - Springfield Clinic LLP, Springfield, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Maine Eye Center, Portland, Maine
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Research Institute at New England Retina Consultants, Springfield, Massachusetts
  - Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Long Island Vitreoretinal Consultants, Hauppauge, New York
  - Asheville Eye Associates - Retina Division, Asheville, North Carolina
  - North Carolina Retina Associates, Cary, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Piedmont Retina Specialists - Winston Salem Office, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Verum Research, LLC, Eugene, Oregon
  - Eyehealth Northwest Portland, Portland, Oregon
  - Cascade Medical Research Institute, Springfield, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Palmetto Retina Center, Aiken, South Carolina
  - ReƟna Consultants of Charleston, Beaufort, South Carolina
  - Charleston Neuroscience Center, Charleston, South Carolina
  - Southeastern Retina, Chattanooga, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Southwest Retina Specialists, Amarillo, Texas
  - Texas Retina Associates- Arlington, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates - Plano, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Tennessee Retina PC, Nashville, Texas
  - Retina Consultants of Texas San Antonio, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Eye Clinic of Wisconsin, Wausau, Wisconsin
- Australia (5):
  - Eye Clinic Albury Wodonga, Albury, New South Wales
  - Strathfield Retina Clinic, Melbourne, New South Wales
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Kepler Universitätsklinikum, Linz
- Canada (4):
  - Calgary Retina Consultants, Calgary, Alberta
  - Alberta Retina Consultants, Edmonton, Alberta
  - Ivey Eye Institute, London, Ontario
  - Retina Centre of Ottawa, Ottawa, Ontario
- Czechia (3):
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Všeobecná fakultní nemocnice V Praze, Prague
  - Axon Clinical, s.r.o. Ocni Klinika, Prague
- France (8):
  - Groupe Hospitalier Pellegrin - CHU de Bordeaux, Bordeaux
  - Service d'Ophtalmologie Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Dijon Bourgogne - Hôpital François Mitterrand, Dijon
  - Centre Ophtalmologique Pôle Vision Val d'Ouest, Écully
  - Centre Monticelli Paradis d'Ophtalmologie, Marseille
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Lariboisière - Service d'ophtalmologie, Paris
  - Centre Ophtalmologique Maison Rouge, Strasbourg
- Germany (5):
  - Dietrich Bonhoeffer Klinikum Klinik für Augenheilkunde, Neubrandenburg, Mecklenburg-Vorpommern
  - Augenzentrum am St. Franziskus-Hospital, Münster, North Rhine-Westphalia
  - Uni-Augenklinik Bonn, Bonn
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Department für Augenheilkunde, Tübingen
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Budapest Retina Associates, Budapest
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen
  - Ganglion Medical Center, Pécs
- Italy (8):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - IRCCS MultiMedica, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione G.B. Bietti Per Lo Sudio E La Ricerca In Oftalmologia - Presidio, Roma
  - Fondazione PTV Policlinico Tor Vergata, Rome
  - Fondazione Policlinico Agostino Gemelli, Rome
- Elisabeth Hospital (ETZ) - location TweeSteden ziekenhuis, Tilburg, Netherlands
- New Zealand (2):
  - Southern Eye Specialists, Christchurch, Canterbury
  - Capital Eye Specialists, Te Aro, Wellington Region
- Poland (5):
  - Oftalmika Sp.Zo.O., Bydgoszcz
  - Centrum Diagnostyki I Mikrochirurgii Oka Lens Sp. Z O.O., Olsztyn
  - Ośrodek Chirurgii Oka Prof. Zagórskiego Sp. Z o.o., Rzeszów
  - Caminomed Sp. Z O.O., Tarnowskie Góry
  - Warszawski Szpital Okulistyczny, Warsaw
- Spain (10):
  - Oftalvist IMED Burjassot, Valencia, Burjasso
  - Institut Català de Retina, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Arruzafa - Metavisión Arruzafa, Córdoba
  - Clínica Baviera, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Universitari General de Catalunya - Grupo Quironsalud, Sant Cugat del Vallès
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (3):
  - Moorfields Eye Hospital NHS foundation Trust, London
  - King's College Hospital, London
  - The Retina Clinic, London

IPD SHARING:
Plan to Share IPD: No